CLINICAL TRIAL: NCT00761228
Title: A Double-blind, Placebo-controlled, Randomized Study of the Safety and Efficacy of NH001 in Improving the Functional Outcome of Patients in a Vegetative State or Minimally Conscious State Following a Severe Traumatic Brain Injury
Brief Title: Efficacy Study of NH001 in Vegetative State & Minimally Conscious State Following a Traumatic Brain Injury
Acronym: NH001-2
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroHealing Pharmaceuticals Inc. (Industry)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3337
Record Dates: First submitted 2008-09-26; First posted 2008-09-29 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Brain Injury
Keywords: Vegetative State; Minimally Conscious State; Coma; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries; Persistent Vegetative State; Coma; Brain Injuries, Traumatic | interventions — Apomorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apomorphine (Active Comparator): Patients will receive an ascending dosing schedule to reach a maximum infusion rate of up to 6 mg/hour for 12 hours a day.
  Interventions: Drug: Apomorphine
- Placebo (Placebo Comparator): Patients will receive a continues subcutaneous infusion of saline solution.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apomorphine — Patients will receive an ascending dosing schedule of continuous subcutaneous apomorphine to reach a maximum infusion rate of up to 6 mg/hour for 12 hours a day.
  Arms: Apomorphine
Drug: Placebo — Patients will receive a continues subcutaneous infusion of saline solution.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the drug apomorphine in subjects who are in a Vegetative State or a Minimally Conscious State.

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized, double-blind, placebo-controlled study of the safety and efficacy of NH001 to improve the functional outcome of patients in a vegetative state or minimally conscious state following a severe traumatic brain injury (TBI).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between 18 and 50 years of age, inclusive.
2. Male or non-pregnant female (females of child-bearing potential will be required to have undergone a pregnancy test with negative results prior to entry to the study).
3. Patients will have sustained a severe closed head injury within one to four months.
4. Patients will have remained in a vegetative or minimally conscious state between one and four months after injury.
5. Patients will have reached a stabilized clinical state prior to admission to the study (e.g. afebrile, haemodynamic and electrolyte stability).
6. Patients will have a mean DRS score between 17 and 29, when measured twice a day over two consecutive days.
7. Informed consent from a legal representative will have been obtained, according to the procedures outlined in Section 8.1.2.
8. Patients who, according to the investigator's opinion, are likely to be available for the required 180-day follow up evaluation.

Exclusion Criteria:

1. Patients who are not clinically stable at the time of entry into the study (infections, cardiovascular decompensation, etc.)
2. Patients who require mechanical respiratory assistance.
3. Patients who show signs of progressive neurological deterioration post-TBI.
4. Patients with a known history of medically relevant substance abuse.
5. Patients with history of cardiac disease.
6. Patients who suffered an anoxic event.
7. Patients who have received an investigational drug within 30 days of the study.
8. Patients who have previously used NH001, other dopaminergic agent (e.g. levodopa, amantadine, domperidone) or any known neuro-stimulant (e.g. methylphenidate, amphetamines, atomoxetine, modafinil) within the last 7 days days.
9. Patients who are receiving dopamine blockers (e.g. risperidone, haloperidol, chlorpromazine, flupenthixol, clozapine, olanzapine, quetiapine)
10. Patients who are receiving drugs of the 5HT3 antagonist class, including, for example, ondansetron, granisetron, dolasetron, palonosetron and alosetron.
11. Patients who are receiving tricyclic antidepressants drugs
12. Patients who are receiving type I antiarrhythmics (i.e. quinidine).
13. Patients who have a known history of cardiac arrhythmias or congenital QTc prolongation.
14. Patients who have a known history of previous neurological functional impairment (e.g. stroke, spinal cord injury, dementia, epilepsy, psychiatric diseases).
15. Patients who experienced seizures within the first week post injury or have ongoing seizures.
16. Patients receiving prophylactic anti-convulsive medications.
17. Patients with known allergies to apomorphine, morphine, sulfites or trimethobenzamide.
18. Patients who are receiving nitrates or other vasodilators.
19. Patients receiving CNS acting agents such as barbiturates, morphine, belladonna, opiates.
20. For male patients, patients who are receiving trazodone or any other drug that is known to produce priapism.
21. Patients without a relative or legal guardian to consent to the study.
22. Patients who, according to the investigator's opinion, are unlikely to be available for the required 180-day follow up evaluation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2010-07; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of meaningful responses to external commands based on Coma Recovery Scale-Revised | Day 42 or the day that the drug treatment is discontinued, whichever happens earlier.

SECONDARY OUTCOMES:
Coma/Near Coma Scale (CNC) Disability Rating Scale (DRS), Glasgow Outcome Scale Extended (GOS-E), ability to participate in 3 hours a day of active rehabilitation, and a clinical impression of change. | Baseline, weekly during drug treatment and at follow up visits of days 90,180 and 360.

CONTACTS AND LOCATIONS:
Overall Officials: Elkan R Gamzu, PhD, Principal Investigator — NeuroHealing Pharmaceuticals Inc.; Ross D Zafonte, DO, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States